CLINICAL TRIAL: NCT01138852
Title: Ampicillin / Sulbactam Versus Cefuroxime as Antimicrobial Prophylaxis for Cesarean Section: a Randomized Study
Brief Title: Ampicillin/Sulbactam Versus Cefuroxime as Antimicrobial Prophylaxis for Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Eleftherios Ziogos, Department of Obstetrics and Gynecology, Nikaia's Regional General Hospital "Agios Panteleimon", Pireaus, Department of Obstetrics and Gynecology, Nikaia's Regional General Hospital "Agios Panteleimon", Pireaus and Department of Infectious Disease Attikon General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UHATpro1
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2004-07

CONDITIONS: Surgical Site Infections
Keywords: post-cesarean infections; ampicillin-sulbactam; cefuroxime; cesarean
MeSH Terms: conditions — Surgical Wound Infection | interventions — sultamicillin; Cefuroxime

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ampicillin-sulbactam (Experimental): This is the drug used to prevent post-cesarean infection
  Interventions: Drug: Ampicillin-sulbactam; Drug: Cefuroxime
- cefuroxime (Active Comparator): This drug was compared to ampicillin sulbactam for prevention of infection
  Interventions: Drug: Ampicillin-sulbactam; Drug: Cefuroxime

INTERVENTIONS:
Drug: Ampicillin-sulbactam — Patients were randomly assigned to receive either 1.5g of cefuroxime, or 3g of ampicillin/ sulbactam intravenously after the time the umbilical cord was clamped
Drug: Cefuroxime — Patients were randomly assigned to receive either 1.5g of cefuroxime, or 3g of ampicillin/ sulbactam intravenously after the time the umbilical cord was clamped

SUMMARY:
The efficacy and safety of a single dose of ampicillin/sulbactam compared to a single dose of cefuroxime at cord clamp for prevention of postcesarean infectious morbidity has not been assessed.

Women scheduled for cesarean delivery were randomized to receive a single dose of either 3g of ampicillin-sulbactam or 1.5g of cefuroxime intravenously, after umbilical cord clamping. An evaluation for development of postoperative infections and risk factor analysis was performed.

DETAILED DESCRIPTION:
The efficacy and safety of a single dose of ampicillin/sulbactam compared to a single dose of cefuroxime at cord clamp for prevention of postcesarean infectious morbidity has not been assessed.

The investigation was designed to evaluate the efficacy and safety of a single dose of ampicillin/sulbactam 3g compared to a single dose of cefuroxime 1.5g in preventing postoperative morbidity. The primary outcome was development of an infection either at the surgical site or elsewhere e.g. urinary tract infection.

A prospective randomized controlled study was performed from July 2004 to December 2008 in one major tertiary care hospital in Athens Greece. All patients undergoing a cesarean delivery were eligible.Patients were randomly assigned to receive either 1.5g of cefuroxime, or 3g of ampicillin/ sulbactam intravenously after the time the umbilical cord was clamped.

ELIGIBILITY:
Inclusion Criteria:

- All patients undergoing a cesarean delivery were eligible.

Exclusion Criteria:

* Patients with known hypersensitivity to penicillin or cephalosporins.
* Patients who required concomitant antibiotic therapy during surgery.
* Patients who have received antibiotics during the 72 hours immediately preceding their enrollment.
* Patients whose postpartum fever was clearly associated with other known causes.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2004-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

REFERENCES:
- [Derived] Williams MJ, Carvalho Ribeiro do Valle C, Gyte GM. Different classes of antibiotics given to women routinely for preventing infection at caesarean section. Cochrane Database Syst Rev. 2021 Mar 4;3(3):CD008726. doi: 10.1002/14651858.CD008726.pub3. PMID 33661539
- [Derived] Ziogos E, Tsiodras S, Matalliotakis I, Giamarellou H, Kanellakopoulou K. Ampicillin/sulbactam versus cefuroxime as antimicrobial prophylaxis for cesarean delivery: a randomized study. BMC Infect Dis. 2010 Nov 30;10:341. doi: 10.1186/1471-2334-10-341. PMID 21118502